CLINICAL TRIAL: NCT05284591
Title: Prospective, Multicenter, Non-interventional Study to Evaluate Patient and Healthcare Provider Satisfaction of Daratumumab Use in the Treatment of First-line Daratumumab, Lenalidomide, Dexamethasone (DRd) Multiple Myeloma Patients as Per Routine Clinical Practice in Germany Depending on Application Route (sc or iv)
Brief Title: Non-interventional Study to Evaluate Patient and Healthcare Provider Satisfaction of Daratumumab Use in the Treatment of First-line Daratumumab, Lenalidomide, Dexamethasone (DRd) Multiple Myeloma Patients in Germany Depending on Application Route (sc or iv)
Acronym: MYLENE
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: 54767414MMY4047
Record Dates: First submitted 2022-02-17; First posted 2022-03-17 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Multiple Myeloma; Newly Diagnosed; Transplant Ineligible; Patient Satisfaction; Patient Preference; Personal Satisfaction
Keywords: Daratumumab; DARZALEX; Lenalidomide; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma; Patient Satisfaction; Patient Preference; Personal Satisfaction | interventions — daratumumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DRd with daratumumab iv de novo: Patients either continue DRd with daratumumab iv, switch to daratumumab sc or switch multiple times iv/sc
  Interventions: Biological: Daratumumab
- DRd with daratumumab sc de novo: Patients either continue DRd with daratumumab sc, switch to daratumumab iv or switch multiple times sc/iv
  Interventions: Biological: Daratumumab

INTERVENTIONS:
Biological: Daratumumab — intravenous or subcutaneous
  Other Names: Darzalex

SUMMARY:
MYLENE is a prospective, multicenter, NIS to evaluate the patient and HCP satisfaction of sc and iv application of daratumumab in routine clinical practice in Germany. Patients observed in this study will be transplant ineligible NDMM patients for which the physician foresees an anti-myeloma therapy using DRd regimen as per local label.

250 NDMM patients treated with DRd will be enrolled (excluding screening failures, i.e., enrolled patients not fulfilling selection criteria identified before treatment start will be replaced) within 12 months in a proportion of approximately 1/3 patients receiving daratumumab sc and 2/3 patients receiving daratumumab iv as per physician's decision.

DETAILED DESCRIPTION:
Therapy options for MM are mainly dependent on the age and fitness of the patients. NDMM patients up to the age of 65-70 years in whom autologous stem cell transplantation is not indicated, anti-myeloma treatment traditionally consists of systemic chemotherapy, with adjunctive use of radiation or surgery in selected cases associated with extramedullary disease. However, the therapeutic landscape of multiple myeloma progressed in the past decade with the introduction of immunomodulatory agents, proteasome inhibitors and anti-CD38 antibodies, like Daratumumab.

After approval of daratumumab iv in May 2016, the sc daratumumab application route was approved in June 2020 in Germany. Real-world evidence data, however, are not yet available neither related to daily experience nor to satisfaction with daratumumab sc application nor to the proportion of patients potentially switching from daratumumab iv to sc application.

MYLENE aims to close these gaps with focus on NDMM patients who are ineligible for autologous stem cell transplantation and who will be treated with DRd; this is to guarantee a homogenous patient population.

All aspects of treatment and clinical management of patients will be in accordance with local clinical practice and applicable local regulations, and at the discretion of the healthcare provider (or treating physician where different). Only data available per clinical practice will be collected within this study. Additionally, where permitted in accordance with local regulations, healthcare providers will be asked to obtain patient-reported outcome (PRO) data from patients within this study. Despite use of PROs and HCP as well as physician questionnaires, the design is non-interventional due to the fact that the questionnaires are structured documentation aids to document questions that are routinely part of the dialog between patient and physician or HCP during the patient visit and/or drug administration or that are considered by the HCP when evaluate treatment for the patient but are not documented in the medical record.

MYLENE is unique as it is focusing on the satisfaction of all involved stakeholders (i.e., patients and HCPs) under real-word conditions and mainly in private practices, since this patient collective is treated preferentially in these institutions, allowing to receive direct feedback about the use of daratumumab sc application and its potential hurdles or/and limitations. Furthermore, this study will provide insights on how the sc/iv application is managed in clinical routine as well as how it is perceived by medical professionals over time.

This NIS will be analyzed exploratively and is hence not designed to confirm or refute a predefined hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Newly diagnosed multiple myeloma (NDMM) and decision for first-line treatment with daratumumab/lenalidomide/dexamethasone (DRd) according to SmPCs of daratumumab
* Each patient must sign an informed consent form (ICF) indicating that he or she understands the purpose of the study and is willing to participate in the study
* Willingness and ability to read, understand and complete patients' questionnaires due to the primary objective of the NIS (i.e., patient satisfaction using the Patient Satisfaction and Time Questionnaire (PatSTQ)).

Exclusion Criteria:

* Participation in an interventional clinical trial (participation in another non-Janssen sponsored NIS or registry is allowed)
* Prior anti-myeloma therapy, with the exception of local radiation therapy or an emergency use of a short course of corticosteroids before treatment
* Any restrictions/limitations preventing to be treated with DRd as per SmPCs of daratumumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MYLENE is focusing on the satisfaction of all involved stakeholders (i.e., patients and HCPs) mainly in private practices, since this patient collective is treated preferentially in these institutions, allowing to receive direct feedback about the use of daratumumab sc application and its potential hurdles or/and limitations.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction and Time with the application route of daratumumab (iv/sc) | For patients with continuous application route the time frame will be 12 months. For patients with switch of application route, at least 4 daratumumab applications after the first switch should be documented.
  The primary objective of this NIS is to exploratively analyze patients' satisfaction of sc and iv application of daratumumab over time as measured by the "Patient Satisfaction and Time Questionnaire" (PatSTQ).
  Overall patients´ satisfaction with daratumumab administration will be displayed as the result of one defined question in the PatSTQ, with descriptive statistics and boxplots.
  Results of PatSTQ will be displayed with frequencies per group and by time point. Additionally, stacked bar plots with questionnaire results (including missings) per item and time point will be presented

SECONDARY OUTCOMES:
HCP satisfaction and time with the application route of daratumumab (iv/sc) | Time frame will be approx. 12 months depending on switch of application route.
  The secondary objective of this NIS is to assess HCPs' satisfaction of sc and iv application over time as measured by the "HCP Satisfaction and Time Questionnaire - patient specific" (HSTQ-ps).
  HCPs' application route satisfaction will be displayed by questionnaire time point as result of the HSTQ - ps questionnaire with frequencies for questions and with descriptive statistics.
Proportion of HCP active time spent on activities | Time frame will be approx. 12 months depending on switch of application route.
  The proportion of HCP active time spent on activities (drug preparation, drug administration, patient care/patient monitoring) over time
Patients' chair time over time | Time frame will be approx. 12 months depending on switch of application route.
  Patients' chair time over time
Patients' overall time spent at doctor's office | Time frame will be approx. 12 months depending on switch of application route.
  Patients' overall time spent at doctor's office
Switch rate (proportion of patients) of daratumumab application routes | Time frame will be approx. 12 months depending on switch of application route.
  The switch rate (proportion of patients) of daratumumab application routes during 12 months of study participation under real-word conditions
Median switch time | Time frame will be approx. 12 months depending on switch of application route.
  Median switch time
Main reasons for sc or iv application selection | Time frame will be from date of site activation (start of potential enrolment at site) to site close-out (up to 14 months after last patient in)..
  The main reasons for sc or iv application selection evaluated by both, the "Physician Therapy Decision Questionnaire - general" (PTDQ-g) at study start and at the end of study (i.e., study close-out) and by the "Physician Therapy Decision Questionnaire - patient specific" (PTDQ-ps) at baseline and at switch of the application route
Impact of different factors on therapy decision and application route selection (PTDQ-ps) | Time frame will be approx. 12 months depending on switch of application route.
  The impact of different factors on therapy decision and application route selection will be displayed as parameter estimates for selected fixed covariates (age, cytogenetics (high vs standard) and relevant comorbidities) in a mixed effects logistic regression model with the result of PTDQ-ps as outcome.
  The treating physician selects up to two main reasons why the (new) application route (sc or iv) of daratumumab for a patient is chosen.
Patients' preference of the application route | Time frame will be approx. 12 months depending on switch of application route.
  Patients' preference of the application route (only for patients switching from one application route to another) as measured by the "Patient Preference Questionnaire" (PatPQ).
  The patient selects which method of daratumumab administration (iv or sc) is preferred and up to two reasons for the preference.

OTHER OUTCOMES:
Safety and tolerability of daratumumab treatment. Occurence and number of patients with adverse events as assessed by CTCAE. | Time frame will be approx. 12 months depending on switch of application route. (On-treatment period: from day of first dose of daratumumab to 30 days after last dose of daratumumab, or end of documentation period, whatever comes first.)
  Occurence and number of patients with (treatment-related) adverse events will be provided.
  Additionally, summary tables of selected subsets of AEs will be displayed summarized by system organ class (SOC) and preferred term (PT), sorted by frequency of SOC and PT. Summary tables for AEs will include only AEs that started or worsened during the on-treatment period. However, safety data from the pre- and post-treatment periods will be listed separately.
  Time to first occurrence of AESI will be calculated for patient with an AESI as the time from the date of first application of daratumumab until onset of first documented AESI and will displayed with descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Knauf, Prof. Dr., Principal Investigator — Centrum für Hämatologie und Onkologie Bethanien, Frankfurt/ Main
Locations (1):
- Centrum für Hämatologie und Onkologie Bethanien, Frankfurt am Main, Hesse, Germany